CLINICAL TRIAL: NCT04696666
Title: Multicenter Clinical Study of the Efficacy and Tolerability of INSTYLAN (Sodium Hyaluronate 80mg/50ml) in Patients With Early or Late Symptoms of Moderate to Severe Hemorrhagic Cystitis Caused by Pelvic Radiation Therapy and/or Chemotherapy
Brief Title: Tolerability and Efficacy of INSTYLAN in Subjects With Moderate to Severe Hemorrhagic Cystitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LIDDE Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-INST01F
Record Dates: First submitted 2021-01-03; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hemorrhagic Cystitis
Keywords: Hemorrhagic cystitis
MeSH Terms: conditions — Cystitis, Hemorrhagic

STUDY DESIGN:
Intervention Model Description: It is a multicenter single-arm clinical study aimed at assessing the efficacy and tolerability of INSTYLAN (Sodium Hyaluronate 80mg/50ml) provided in routine clinical practice in patients presenting with symptoms of moderate to severe hemorrhagic cystitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients assigned in a single group and treated with 6 instillations of INSTYLAN for 6 weeks (Experimental): Single Group Assignment
  Interventions: Device: INSTYLAN (Sodium Hyaluronate 80mg/50ml)

INTERVENTIONS:
Device: INSTYLAN (Sodium Hyaluronate 80mg/50ml) — The bladder instillation with INSTYLAN is a treatment involving a sterile solution of Sodium Hyaluronate (80mg/50ml) inserted into the bladder through a catheter and released after a short period of time.

SUMMARY:
The purpose of this study is to assess the efficacy and tolerability of INSTYLAN (Sodium Hyaluronate 80mg/50ml) in Patients with early or late symptoms of moderate to severe hemorrhagic cystitis caused by pelvic radiation therapy and/or chemotherapy. The study is conducted in the field of routine clinical practice and will recruit 30 subjects treated with intravesical instillations with INSTYLAN weekly for 6 weeks.

DETAILED DESCRIPTION:
This is a multicenter single-arm clinical study including male and female subjects with moderate to severe hemorrhagic cystitis caused by pelvic radiation therapy and/or chemotherapy as determined by the physician. A total of 30 subjects are anticipated and will be enrolled in 10 study sites in France.

The patients will receive intravesical instillations with INSTYLAN weekly for 6 weeks.

The objectives of the study are to assess the efficacy of intravesical instillations of INSTYLAN on the basis of hemorrhagic cystitis symptoms disappearance. The primary endpoint is the evaluation of pain using a verbal rating scale one week and four weeks after treatment versus Baseline.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, at least 18 years,
* Patients who provided signed written informed consent, which includes compliance with requirements listed in the consent form,
* Patients with diagnosis of Hemorrhagic Cystitis,
* Patients with diagnosis of bladder pain (pressure or pelvic discomfort) with at least one other urinary symptom (need to urinate right away (urgency), often (frequency), or both).

Exclusion Criteria:

* Patients with Post-void residual (PVR) urine volume > 200ml,
* Patients presently treated with intravesical treatment (replenishment therapy with glycosaminoglycans),
* Patients receiving HyperBaric Oxygen Therapy (HBOT),
* Patients with neurogenic bladder,
* Patients treated with neuromodulation techniques within the last six months,
* Patients undergoing or scheduled for radiation therapy, brachytherapy, chemotherapy or treatment with BCG or with Mitomycin-C,
* Patients suffering from lower urinary infections (UTIs),
* Patients with unstable cardiovascular disease,
* Patients with any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in the intensity of bladder pain from the beginning of the study (baseline: Week 1) to Week 7 | Week 7
  Questionnaire with 5 closed-ended response options: no pain, slight pain, moderate pain, severe pain, very severe pain
Change in the intensity of bladder pain from the beginning of the study (baseline: Week 1) to Week 10 | Week 10
  Questionnaire with 5 closed-ended response options: no pain, slight pain, moderate pain, severe pain, very severe pain

SECONDARY OUTCOMES:
Evaluation of hematuria following a rating scale | Baseline, week 7 and week 10
  Verbal rating scale of the colour of the urines: yellow, pink or red-brownish
Evaluation of number of micturitions / 24 hours | Baseline, week 7 and week 10
  Voiding diary sheet for each 24-hour period
Evaluation of urgency of micturitions following a rating scale | Baseline, week 7 and week 10
  Verbal rating scale (slight, moderate, important)

CONTACTS AND LOCATIONS:
Overall Officials: Marc FOURMARIER, MD, Principal Investigator — Aix en Provence Hospital Center (Aix en Provence)
Locations (10):
- France (10):
  - Aix en Provence Hospital Center, Aix-en-Provence
  - Ajaccio Hospital Center (Notre Dame de la Miséricorde), Ajaccio
  - Polyclinic Sainte Marguerite (Auxerre), Auxerre
  - Clinic Rhône Durance (Avignon), Avignon
  - Cahors Hospital Center, Cahors
  - Clinic of Val d'Ouest (Ecully), Écully
  - Mutualist Clinic Porte de l'Orient (Lorient), Lorient
  - Clinic Saint George (Nice), Nice
  - Saint Louis University Hospital Center (Paris), Paris
  - Regional University Hospital Center (Strasbourg), Strasbourg